CLINICAL TRIAL: NCT02085915
Title: Evaluation of the Strip PeriScreen for the Fast Diagnosis of the Spontaneous Infection of the Liquid of Ascites During the Cirrhosis
Acronym: Per-DRISLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHD 065-13
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Cirrhosis; Liquid of Ascites; Infection
MeSH Terms: conditions — Fibrosis; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- strip Peri Screen (Other)
  Interventions: Other: strip Peri Screen

INTERVENTIONS:
Other: strip Peri Screen

SUMMARY:
The forecast of the spontaneous infection of the liquid of ascites (ISLA) at the cirrhotic patient is still burdened by a heavy mortality. The fast diagnosis of the ISLA is thus an essential stake to improve the forecast.

Investigators would so like to estimate the interest of the strip PeriScreen for the fast diagnosis of the ISLA at cirrhotic patients . Investigators plan to include 670 patients, what would allow to make out a will at least on ascites 2000 on about twenty centers for duration estimated of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years
* Presence of ascites due to cirrhosis
* Hospitalization for a complication of cirrhosis (ascites first decompensation, gastrointestinal bleeding, encephalopathy, etc ...).

or

* Hospitalization to perform a paracentesis evacuated outpatient
* Patients on long-term antibiotic primary or secondary prophylaxis the spontaneous bacterial peritonitis and with clinical and/or biological signs that suggest spontaneous infection of ascite.

Exclusion Criteria:

* Patients with ascites urgently admitted to hospital for suspected infection receiving antibiotics for more than 12 hours.
* chylous ascites,
* Hemorrhagic Ascites
* Biliary Ascites (straw)
* Ascites heterogeneous appearance
* Ascites not related to portal hypertension (peritoneal carcinomatosis, pancreatic ascites, tuberculosis, etc ...)
* Patient receiving imipenem IV.
* Patients on long-term antibiotic primary or secondary prophylaxis the spontaneous bacterial peritonitis without clinical and/or biological signs that suggest spontaneous infection of ascite.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
liquid of ascites spontaneous infection | Baseline
  Periscreen strip compared to the cytological analysis

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu SCHNEE, Dr, Study Director — CHD Vendée La Roche sur Yon
Locations (22):
- Hopital Jolimont, Haine-Saint-Paul, Belgium
- France (21):
  - CH Amiens, Amiens
  - CHU Besançon, Besançon
  - CHRU de Brest, Brest
  - CH Caen, Caen
  - CH Cholet, Cholet
  - Hopîtal Beaujon, Clichy
  - Hopital Laennec, Creil
  - CH Dijon, Dijon
  - CH Gonesse, Gonesse
  - CHD Vendée, La Roche-sur-Yon
  - CH Lille, Lille
  - CHU Nice, Nice
  - CH Orléans, Orléans
  - CH Reims, Reims
  - CH Rennes, Rennes
  - CH Rouen, Rouen
  - CH St Antoine, Saint-Antoine
  - CH Yves Le Foll, Saint-Brieuc
  - CH Saint-Denis - Hôpital de la Fontaine, Saint-Denis
  - Hôpital Purpan, Toulouse
  - CH Vannes, Vannes